CLINICAL TRIAL: NCT06102200
Title: Prisma Health Clemson University
Brief Title: An Integrated Intervention Involving Recovery Coaching and Cognitive Behavioral Therapy for Opioid Use Disorder
Acronym: OVERCOME 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1930664-6; R34DA057662 (NIH)
Record Dates: First submitted 2023-08-31; First posted 2023-10-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Standard of Care; Standard of Care + CBT4CBT; Standard of Care + CBT4CBT + RC
Keywords: CBT; Peer recovery coach; Opioid

STUDY DESIGN:
Intervention Model Description: Behavioral intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care (Active Comparator): Participants in the standard of care condition will receive the standard treatment at the recovery program, which consists of weekly, bi-weekly or monthly visits (at the discretion of the provider) in-person or virtually. This condition will be matched with the other conditions in terms of the number of research visits.
  Interventions: Behavioral: Sandard of care
- Standard of care + CBT4CBT (Experimental): This condition will integrate the standard of care and CBT4CBT interventions. The CBT4CBT is an 8-session (module) system for teaching with one module on the basics of buprenorphine and the other modules on the seven CBT core skills tailored around issues related to buprenorphine and OUD and other SUDs: (1) Introduction to functional analysis of substance use; (2) strategies for recognizing and coping with craving; (3) refusal skills and assertiveness; (4) training in problem-solving skills; (5) strategies for recognizing and changing thoughts; (6) decision-making skills; (7) how to use CBT skills to reduce HIV/ HCV risk. Each module takes 30 minutes to complete and has a format, which includes on-screen narration, animation, quizzes, and interactive exercises to teach and model effective use of skills. Modules end with a practice exercise.
  Interventions: Behavioral: CBT4CBT
- Standard of care + CBT4CBT+ RC (Experimental): This condition will integrate the standard of care, CBT4CBT, and recovery coaching services with Assertive Community Engagement (ACE) model interventions. The CBT4CBT is an 8-session (module) system for teaching with one module on the basics of buprenorphine and the other modules on the seven CBT core skills tailored around issues related to buprenorphine and OUD and other SUDs Peer recovery coaching services involve a form of nonclinical, peer support aimed at helping individuals with substance use disorders to achieve and maintain recovery. Recovery coaches are individuals with experience with substance use and successful recovery. In addition to their lived experience, recovery coaches obtain formal training on substance use coaching and receive ongoing supervision. The recovery coaches use an assertive engagement approach to provide holistic, person-centered, and strength-based support.
  Interventions: Behavioral: CBT4CBT; Behavioral: RC

INTERVENTIONS:
Behavioral: CBT4CBT — This condition will integrate the standard of care and CBT4CBT interventions. The CBT4CBT is an 8-session (module) system for teaching with one module on the basics of buprenorphine and the other modules on the seven CBT core skills tailored around issues related to buprenorphine and OUD and other SUDs: (1) Introduction to functional analysis of substance use; (2) strategies for recognizing and coping with craving; (3) refusal skills and assertiveness; (4) training in problem-solving skills; (5) strategies for recognizing and changing thoughts; (6) decision-making skills; (7) how to use CBT skills to reduce HIV/ HCV risk. Each module takes 30 minutes to complete and has a format, which includes on-screen narration, animation, quizzes, and interactive exercises to teach and model effective use of skills. Modules end with a practice exercise.
  Other Names: CBT4CBT-Buprenorphine
  Arms: Standard of care + CBT4CBT; Standard of care + CBT4CBT+ RC
Behavioral: RC — Peer recovery coaching services involve a form of nonclinical, peer support aimed at helping individuals with substance use disorders to achieve and maintain recovery. Recovery coaches are individuals with experience with substance use and successful recovery. In addition to their lived experience, recovery coaches obtain formal training on substance use coaching and receive ongoing supervision. The recovery coaches use an assertive engagement approach to provide holistic, person-centered, and strength-based support.
  Other Names: Recovery Coaching
  Arms: Standard of care + CBT4CBT+ RC
Behavioral: Sandard of care — Participants in the standard of care condition will receive the standard treatment at the recovery program, which consists of weekly, bi-weekly or monthly visits (at the discretion of the provider) in-person or virtually. This condition will be matched with the other conditions in terms of the number of research visits.
  Arms: Standard of care

SUMMARY:
The Overcome II study is a randomized controlled trial among adults receiving sublingual buprenorphine to help prevent or reduce illicit drug use. The study outcomes will be compared between three treatment arms: (1) sublingual buprenorphine only, which is the standard-of-treatment (2) sublingual buprenorphine with a computer-based cognitive behavior therapy for substance use disorders (CBT4CBT), (3) sublingual buprenorphine with CBT4CBT and peer recovery coaching. The primary outcome of interest is the reduction in the proportion of positive results for saliva toxicology screenings for any drug during the 8-week treatment period. Study participants will also be assessed for the outcomes of retention to standard-of-treatment and illicit drug use at 1-, 3-, and 6-months follow-ups after the end of treatment.

DETAILED DESCRIPTION:
Buprenorphine has proven to be an effective pharmacologic strategy for treating OUD. However, buprenorphine is unlikely to give greater overall protection because of the shorter duration of treatment. There is a need for studies on interventions that could increase retention to buprenorphine, especially among those with ongoing illicit substance and polysubstance use.

Using a randomized controlled trial study design, the Overcome II study aims to investigate the incremental benefit in terms of reduction in illicit drug use and retention in standard of treatment due to providing the peer recovery coach and/or CBT4CBT interventions as a compliment to standard-of-treatment among persons receiving medication for opioid use. The study outcomes will be compared between three treatment arms: (1) sublingual buprenorphine only, which is the standard-of-treatment (2) sublingual buprenorphine with CBT4CBT, (3) sublingual buprenorphine with CBT4CBT and peer recovery coaching. The primary outcome of interest is reduction in the proportion of positive results for saliva toxicology screenings for any drug during the 8-week treatment period. Study participants will also be assessed for the outcomes of retention to standard-of-treatment and illicit drug use at 1-, 3-, and 6-months follow-ups after the end of treatment. The institutional review board at Prisma Health will provide the oversight for the ethical conduct of the study. Potential participants at Prisma Health will be screened for eligibility, will undergo the informed consent procedure, and eligible persons who consent to participation will be recruited into the study.

The participants will be randomized of one of the three treatment arms in a 1:1:1 ratio. The study will aim to recruit 30 participants per treatment arm. Study procedures will be conducted both virtually and at research facilities of the Prisma Health Addiction Medicine Center, in Greenville, SC. Participants will attend the research visits once a week during the first eight weeks (sessions 1 to 8), and 1-, 3-, and 6- months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age);
2. DSM-V diagnosis of OUD, confirmed via electronic medical record review;
3. Currently receiving SL buprenorphine/ naloxone and/or buprenorphine HCL;
4. Initiated SL buprenorphine within the last 30 days;
5. Willing to accept a random assignment to either treatment arm:
6. Adequate computer skills

Exclusion Criteria:

1. Severe medical or psychiatric disability that could impair the ability to perform study related activities (determined by the clinician);
2. Pregnancy, planning conception, or breast-feeding for female participants;
3. Inability to independently read and/or comprehend the consent form or other study materials;
4. Inability to read/speak English (inability to independently read and comprehend the consent form or other study materials);
5. Current suicidal ideation based on the Patient Health Questionnaire-9
6. Have taken or received any prescribed buprenorphine product within 30 days prior to the current treatment episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Drug use | 8 weeks
  The percentage of of saliva toxicology screens positive for all drugs during the 8 initial study weeks

SECONDARY OUTCOMES:
Buprenorphine retention at 3-month follow-up | 20 weeks
  Retention to buprenorphine
Buprenorphine retention at 6-month follow-up | 32 weeks
  Retention to buprenorphine
Drug use | 12 weeks
  The percentage of saliva toxicology screens positive for all drugs at 1 month follow-up
Drug use | 20 weeks
  The percentage of saliva toxicology screens positive for all drugs at 3 month follow-up
Drug use | 32 weeks
  The percentage of saliva toxicology screens positive for all drugs at 6 month follow-up
Opioid use | 8 weeks
  The percentage of saliva toxicology screens positive for opioids during the 8 initial study weeks
Opioid use | 12 weeks
  The percentage of saliva toxicology screens positive for opioids at 1 month follow-up
Opioid use | 20 weeks
  The percentage of saliva toxicology screens positive for opioids at 3- month follow-up
Opioid use | 32 weeks
  The percentage of saliva toxicology screens positive for opioids at 6- month follow-up
Self-report drug use | 8 weeks
  Self-report drug use in the past 30 days (yes/no)
Self-report drug use | 12 weeks
  Self-report drug use in the past 30 days (yes/no)
Self-report drug use | 20 weeks
  Self-report drug use in the past 30 days (yes/no)
Self-report drug use | 32 weeks
  Self-report drug use in the past 30 days (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Alain H Litwin, MD, Principal Investigator — Prisma Health
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pericot-Valverde I, Perez A, Heo M, Coleman A, Ortiz E, Merchant K, Melling T, Litwin A. Rationale, design, and methodology of a randomized pilot trial of an integrated intervention combining computerized behavioral therapy and recovery coaching for people with opioid use disorder: The OVERCOME study. Contemp Clin Trials Commun. 2022 May 5;28:100918. doi: 10.1016/j.conctc.2022.100918. eCollection 2022 Aug. PMID 35573387
- [Derived] Pericot-Valverde I, Heo M, Byrne KA, Karasz A, Perez A, Lopes S, Groome M, Voss S, King A, Barnick K, Litwin AH. Rationale and design of a three-arm randomized clinical trial to improve drug use and retention in care of people with opioid use disorder on buprenorphine: OVERCOME II study. Contemp Clin Trials. 2026 Jan 17:108226. doi: 10.1016/j.cct.2026.108226. Online ahead of print. PMID 41554331